CLINICAL TRIAL: NCT06680765
Title: An Evaluation of the Effectiveness of a Maternal, Neonatal and Child Health Component for the Matasa Matan Arewa and Smart Start Interventions Targeting Married Adolescent Girls in Nigeria and Ethiopia
Brief Title: An Evaluation of the Effectiveness of a Maternal, Neonatal and Child Health Component for Matasa Matan Arewa and Smart Start Targeting Married Adolescent Girls in Nigeria and Ethiopia
Acronym: MNCH NG-ET
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Population Services International (Other)
Responsible Party: Principal Investigator, Abednego Musau, Senior Research and Learning Lead - A360, Population Services International
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1735-2023
Record Dates: First submitted 2024-11-07; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Pre-conceptual Care; Antenatal Care; Postpartum Family Planning; Adolescent Maternal Health
Keywords: Health pregnancies; Antenatal care; Pre-conceptual care; Maternal, neonatal and child health; Post-partum family planning
MeSH Terms: interventions — Methylmalonic Acid

STUDY DESIGN:
Intervention Model Description: The study constitutes of an intervention and a comparison group. In Nigeria, the intervention group participants are drawn from the specific LGAs where the MMA program enhanced with the MNCH component is implemented. The comparison group is drawn from LGAs implementing MMA without the MNCH component. The study is conducted in specific PHCs purposely selected to host the evaluation and the catchment areas that are served by the PHCs. In Ethiopia, the study will be implemented in four out of the five regions that implement the Smart Start interventions. The intervention group is drawn from eight (8) woredas in the four regions where Smart Start with Smart pathways is implemented. The comparison group is based in 8 woredas geographically distant from those offering Smart Pathways.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparison group (Active Comparator): Smart Smart and MMA are implemented in primary health centres and health posts by community health nurses, health extension workers or midwives. AGYW undergo counselling as individuals or as a group (for Nigeria through life, family and health classes- four sessions with 15-20 girls). Sessions focus on creating relevance of contraceptives as a tool for pursuing life aspirations and as a means to contribute to the household financial security through birth spacing. Girls who opt to voluntarily adopt modern contraceptive methods receive them on spot or at a later date based on their preferences and needs. For Nigeria, sessions are moderated by trained female mentors, while for Ethiopia health extension workers moderate sessions guided by a goal card.
  Interventions: Behavioral: Comparison group
- Intervention group (Experimental): Smart Pathways and MMA plus are the MNCH components which are implemented alongside the respective sexual and reproductive health interventions. These interventions target AGYW (15-19 in Nigeria and 15-24 in Ethiopia). These interventions are implemented at primary health centres and health posts. Eligible women are recruited using a targeted mobilization approach by trained mobilisers. In both locations, AGYW go through sessions covering preconceptual care and nutrition, ANC education and services and referral. Intervention components are delivered by trained health providers at the health centres and posts.
  Interventions: Behavioral: Intervention group

INTERVENTIONS:
Behavioral: Intervention group — These are behavioural interventions delivered by trained HEWs or Health providers at primary care facilities (PHCs in Nigeria and Health posts in Ethiopia).
  Other Names: Smart Pathways and MMA plus
  Arms: Intervention group
Behavioral: Comparison group — These are behavioural interventions delivered by trained HEWs or Health providers at primary care facilities (PHCs in Nigeria and Health posts in Ethiopia).
  Other Names: Smart Start and MMA
  Arms: Comparison group

SUMMARY:
Evidence on the effectiveness of interventions aimed at creating demand and access to pre-conceptual and antenatal care (ANC) among adolescent girls and young women (AGYW) from sub-Saharan Africa is scarce. A program called Adolescents 360 (A360) led by Population Services International in Nigeria, Ethiopia, Kenya and Tanzania supports adolescent girls to identify contraceptives as a relevant tool for enabling them to pursue their self-defined life aspirations. Avoiding or delaying childbirth is crucial for AGYW to pursue their life goals, but motherhood remains a vital aspiration for many. A360 respects these aspirations and supports AGYW to pursue motherhood when the time comes, safely and aligning with their unique preferences. In 2022, A360 set out to design a maternal, neonatal and child health (MNCH) component that would be layered to the existing sexual and reproductive health interventions in Ethiopia and Nigeria. A360 employed human-centered design (HCD) to design these components. The implementation of these components in real-world settings began in 2023. A360 has designed an evaluation to determine the effectiveness of the MNCH components in improving the AGYW's comprehensive knowledge of what is needed to pursue healthy pregnancies, increase their self-efficacy to access ANC and garner support from their key influencers in the process of pursuing healthy pregnancies. The evaluation's primary objective is to determine the effectiveness of the MNCH components at increasing comprehensive knowledge, self-efficacy and key influencer support to pursue healthy pregnancies among married AGYW in Nigeria and Ethiopia. The secondary objectives are: (a) to evaluate the component's effectiveness at increasing comprehensive knowledge of what care is required to attain healthy pregnancies, (b) to evaluate the component's effectiveness at increasing self-efficacy to attend ANC, (c) to determine the component's efficacy at eliciting support from AGYW's key influencers when they are pursuing healthy pregnancies, and (d) to surface the system-level barriers, facilitators, and opportunities for program improvement during the implementation of the MNCH components. The MNCH components are implemented in Kaduna and Jigawa states in Nigeria and in Oromia, Sidama, Amhara, South and Central regions in Ethiopia. The evaluation is based in the same geographies where the components are implemented. The evaluation uses an implementation-effectiveness hybrid design, blending an outcome evaluation and an implementation science component. The outcome evaluation constitutes of a quantitative survey using a longitudinal approach with two study arms, an intervention, and a comparison arm. It has three assessments: a recruitment phase, and two follow-ups (3 months after recruitment and 8 weeks post-partum (only for pregnant AGYW).

Participant recruitment is conducted using recruitment scripts after obtaining oral consent and the administration of a set of screening questions to assess eligibility. Full consenting procedures are executed and written consent obtained prior to involvement in any of the evaluation components. A structured questionnaire is used to gather quantitative data from the survey using a Computer Assisted Personal Interview (CAPI) approach. Furthermore, FGD, IDI and KII facilitation guides are used to gather qualitative data. During this process, all sessions are audio-recorded. Audio records are transcribed verbatim and translated. Data is collected by trained enumerators and qualitative researchers who are certified to conduct human subjects' research. Analysis of quantitative data will follow a repeated measures approach employing generalized estimating equations. The repeated measurements of each subject will be made at two times. Between group t-tests and chi-square tests of comparison will be conducted to identify secondary outcomes which show statistically significant differences between participants in the intervention and comparison arms. The qualitative data transcripts will be rigorously analyzed using NVivo or Dedoose. Open-coding and closed-coding will be utilized to identify themes in the qualitative data. Claim statements attributing change to key intervention drivers will be drawn from narrative stories of program beneficiaries guided by the intervention's theory of change.

The evaluation received ethical approvals from Ethiopian Midwives Association (EMwA) Institutional Review Commitee (IRC) and the PSI Research Ethics Board (REB) prior to the enumerators training and field data collection. Subsequently, the ethical approval letters were submitted to the sub-national health departments for their reference and support in the management of the field work.

DETAILED DESCRIPTION:
Pregnancy and childbirth are a leading cause of morbidity and mortality among adolescent girls. In 2021, maternal conditions were the fourth leading cause of disability-adjusted life years and the second leading cause of mortality among adolescent girls 15-19. The negative health consequences of teen pregnancies include pregnancy complications (pre-eclampsia, unsafe abortion, anaemia, maternal depression), birth complications (pre-term birth, obstructed labour, obstetric fistula), post-partum complications (post-partum haemorrhage, puerperal sepsis, neonatal death, low birth weight neonates and postpartum depression) and death. Further, pregnancy at adolescence is associated with multiple socio-economic outcomes such as discrimination, rejection, social isolation, school discontinuation and economic deprivation. Despite the need to careful monitoring and care needed during pregnancy, most pregnant girls receive poor health care. Fewer pregnant girls, compared to their older counterparts, initiate ANC, attend the recommended number of ANC visits, receive high quality ANC care, are supervised during birth by a skilled health worker or receive postpartum care. There is growing global attention for health systems to make strategic investments to avert teen pregnancies and to deliver high quality, user-friendly and timely interventions for the adolescent girls who conceive.

Motherhood is a key aspiration for most women including those in adolescence. In patriarchal societies, where early marriage is common, girls are expected to begin childbearing immediately after their marriage to prove their fertility. At this age, married adolescent girls lack comprehensive knowledge about pregnancy and childbirth, and have limited agency and decision-making power to determine what is the best care for them. Delivering high quality and timely antenatal care is a crucial intervention that could avert most of the risks associated with adolescent pregnancy. Initiating ANC in early pregnancy provides health workers an opportunity to perform health promotion and education, conduct risk assessment and action, and monitoring and timely management of pregnancy complications. Yet ANC outcomes for pregnant adolescents are wanting. Studies have documented various reasons why ANC attendance is poor for adolescent girls which include health system factors such as the tense relationships with providers, the poor service quality, and long distances to health facilities; social factors such as level of support from the male partner and community norms; and individual factors such as age, level of education, autonomy, knowledge of the importance of ANC, place of residence, financial factors, pregnancy disclosure, parity and marital status. Holistically addressing the factors influencing the timing, consistency and completeness of ANC attendance and improving the quality and user-centredness of ANC for adolescent girls using a socio-ecological model could improve the pregnancy outcomes among pregnant teens and reduce the avoidable complications.

Several interventions have been trialed to increase demand for, utilization and completion of ANC among adolescent girls who are pregnant. These include group ANC and home visits by community health workers. Findings from these studies has shown a promising outlook on the interventions' ability to increase ANC adherence, reduce the gestational age at first ANC attendance, improve the satisfaction with ANC services and skilled attendance at birth. Yet not all expected outcomes from these interventions were attained and only two of the five studies in a systematic review of interventions to increase ANC adherence showed positive results. Group ANC has shown good results at increasing the awareness of at least three pregnancy danger signs among pregnant adolescent girls. In a separate study conducted in Kenya, nutritional and health knowledge relevant to pregnant women were not substantially different between ANC and non-ANC attendees. In a similar study in Tanzania, only 40.2% of women were knowledgeable on the danger signs of pregnancy. A study in Indonesia demonstrated good results of a trial to increasing knowledge across the pregnancy continuum.

Although intervening to increase demand and timeliness of initiating ANC, doing so in the pre-conceptual period, when girls and their partners are considering conceiving offers the most opportune window to create awareness of what things they need to do to attain a healthy pregnancy. This would include what health issues can affect fertility, the desired nutritional behaviors and the signs and symptoms of pregnancy. This would also alert the couple on what things are expected in early pregnancy including access to early ANC. Intervening prior to conception is important, because it provides health workers an opportunity to screen health risks that could prevent conception, but also those which could negatively affect pregnancy outcomes. Despite the recognition of the value of pre-conceptual interventions, there is huge gap of evidence on what interventions would work for adolescent girls at risk of pregnancy to increase demand of and relevance of ANC. First, interventions in this period are less prioritized by health systems and providers. Second, when such interventions exist, they vary widely between geographies with very few of these in developing countries and interventions not being tailored to the needs of adolescent girls. This was affirmed by a scoping review conducted in 2017 which demonstrated that only 6 of the 27 studies on preconceptual interventions were conducted outside of the United States, only one in Lebanon. Although, most of the interventions demonstrated improvement in preconceptual knowledge, change in dietary habits and use of folic acid, none of the studies tracked the impact of the interventions on ANC outcomes, when pregnancy occurred.

The lack of adolescent-specific evidence and the recognition of the number of teen pregnancies in sub-Saharan Africa, does present a valid opportunity for programmers to design, implement and evaluate pre-conceptual and early pregnancy interventions to document their impact on ANC, maternal and neonatal and post-partum outcomes. Since 2016, Population Services International (PSI) and its consortium partners employed human centred design (HCD) techniques to design a user-centered intervention MNCH component targeting married adolescent girls in northern Nigeria and Ethiopia under the Adolescents 360 (A360) project. This component is layered on two signature aspirational sexual and reproductive health interventions, Smart Start for Ethiopia and Matasa Matan Arewa (MMA) for northern Nigeria. The interventions increase demand for and uptake for voluntary modern methods of contraception and counselling services in primary care outlets among married adolescent girls. The MNCH component targets adolescent girls and young women (AGYW) at risk of pregnancy, those actively trying to conceive and those in early pregnancy. The MNCH component for northern Nigeria is called MMA Plus and that in Ethiopia is called Smart Pathways. MMA plus is implemented through Society for Family Health and is implemented through primary care centres (PHCs) in Kaduna and Jigawa states. At the PHCs girls receive services directly through a trained youth-friendly provider and participate in life, family and health (LFH) classes. LFH consists of four guided mentorship sessions conducted over a four-week duration convened by trained mentors. During these sessions girls receive information including nutrition, child spacing, interpersonal communication, financial management and gains life and vocational skills). The MNCH component is built on the LFH classes. Girls who are at risk of pregnancy and who don't want to use a method of contraception or who suspect that they are pregnant are mobilized by female mentors or through their husbands to attend LFH sessions at PHCs. Those who walk in to receive services are offered the services directly and introduced to the LFH classes. The sessions take two hours, are moderated by trained female mentors and attended by ANC experts (trained providers) who offer information and counselling on attaining health pregnancies. Girls who test positive for pregnancy undergo routine ANC, enhanced with gestational age-specific messages about the expectations of ANC, birth preparedness, nutrition during pregnancy, danger signs and how to avoid them and postpartum family planning (PPFP).

In Ethiopia Smart Pathways is layered on Smart Start. Smart Start targets married adolescent girls 15-19 and their spouses. Smart Start is implemented as part of the national Health Extension Program (HEP) through health posts. Health extension workers (HEWs) engage married adolescent girls alone or with their husbands to discuss how the use of modern contraceptive methods to plan their families can facilitate financial planning and enhance the financial security of their families using a Smart Start Counselling guide called a 'goal card'. Smart Pathways targets AGYW 15-24. A team of trained Ministry of Health-recognized community mobilizers consisting of members of the women development army (WDA) approach married adolescent girls from their communities and introduce them to Smart Start. Married AGYW who express interest to take up birth spacing are linked to HEWs who are working in the community or at health posts to receive the Smart Start intervention (pathway 1). AGYW who are ambivalent to receiving contraceptive counselling and services or those who intend to conceive soon are linked by trained mobilizers to a HEW who takes them through the Smart Pathways component for non- pregnant girls. The HEW uses the Smart Pathways guide to discuss issues related to Preconception Care Counselling and early ANC initiation (pathway 2). For AGYW who have missed their periods or suspect they are pregnant, the trained mobilizers link them to health centres or health posts where HEWs or midwives take them through a seven-step process that covers pregnancy testing, building demand for ANC, the benefits and components of ANC, danger signs of pregnancy, smart nutrition, preparation for delivery and post-partum family planning (pathway 3). Girls in Pathway 2 who conceive are referred to navigate through pathway 3 when that time comes. When pregnant AGYW navigate through ANC, they are offered services based on the Ethiopia Federal Ministry of Health antenatal care guidelines (Ministry of Health of Ethiopia, 2022).

Our evaluation employs mixed methods to document the outcomes of the intervention and uncover implementation barriers, facilitators, and opportunities for institutionalization within existing health systems. The main objective is to determine the effectiveness of MNCH intervention components leveraged on existing A360 interventions at increasing comprehensive knowledge, self-efficacy and key influencer support to pursue healthy pregnancies among married AGYW in Nigeria and Ethiopia. The evaluation uses an effectiveness-implementation hybrid study design so that we are able to evaluate the impact of the intervention in real-world settings (i.e., effectiveness) and to assess best approaches to implement the intervention (implementation research). This approach has been established to accelerate the translation of evidence into practice and to increase the usefulness and relevance of research findings for policy decisions. The hybrid design employs mixed methods consisting of a quantitative survey, routinely collected program data and qualitative data. For the implementation research element, the qualitative impact protocol (QuIP) approach is employed alongside traditional qualitative methodologies. Independent qualitative researchers who are not familiar with the interventions' theory of change or who have limited knowledge of the expected changes from the intervention perform exploratory interviews with the beneficiaries will document change stories highlighting what might have contributed to the most significant change in their lives. This reduces the bias associated with an inquiry that focuses on the change specifically brought about by the intervention where beneficiaries might intentionally or unintentionally attribute change to an intervention even when those changes were caused by other factors. This approach involves the use of open-ended and exploratory tools starting with the expected changes and rolling back to associate these with activities that were happening prior to the evaluation. The QuIP methodology is conducted parallel to the quantitative survey and routinely collected program data to triangulate the findings.

This study constitutes of an intervention and a comparison group. In Nigeria the study is based in two states i.e., Kaduna and Jigawa. For the intervention group, the study is conducted in the specific local government areas (LGAs) where the MMA program enhanced with the MNCH component is implemented. For the comparison group, the study is conducted in LGAs implementing MMA without the MNCH component. At the LGAs, the study is conducted in specific PHCs which have been purposely selected to host the evaluation and the catchment areas that are served by the PHCs. In Ethiopia, the study is implemented in five regions implementing Smart Start. The intervention group is drawn from eight (8) woredas in the four regions where Smart pathways is implemented. The comparison group is drawn from 8 woredas geographically distant from those offering Smart pathways but offering Smart Start. The evaluation is conducted in health centres and health posts that offer comprehensive ANC services.

The primary participants for the study are married AGYW aged 15-19 years from Nigeria and 15-24 years in Ethiopia. The study involves a mix of married AGYW who have both experienced a prior pregnancy and those who have not (but at risk of pregnancy). The secondary target groups are (a) male partners (husbands) of married AGYW who have received the MNCH intervention in Nigeria, (b) health providers and community health mobilizers from the intervention locations. For the recruitment of participants, the quantitative survey leverages already existing trained mobilizers to perform recruitment procedures. The mobilizers are trained to identify and recruit AGYW from the community guided by a recruitment script. The mobilizers are familiar with their communities and will approach potential participants directly by face-to-face contact during their routine household visits, in clinics and/or during community gatherings. for the qualitative component participants are recruited primarily through Smart Start and MMA program staff, particularly health extension workers and health providers working at the facilities implementing the MNCH component. The recruiters will be provided with guidance on who should be recruited for focus group discussions (FGDs) and in-depth interviews (IDIs).

The study sample size is 2420 survey participants, 1330 for Ethiopia and 1090 participants in Nigeria. The qualitative component involves four (4) FGDs for each country, 24 IDIs with AGYW, 10 IDIs will husbands and 35 key informant interviews (KIIs) with health providers and mobilisers.

The quantitative data is gathered using a Computer Assisted Personal Interview (CAPI) approach through Survey CTO software. The survey tool is designed in English and local languages of the study regions with a drag and drop user interface. When building the tool in Survey CTO software automated live data checks, extensive validations and cross-checks are programmed. This reduces errors and inaccuracies during the personal interview. The data is synchronized with a web-based server intermittently. The IDIs, FGDs and KIIs are recorded using digital voice recorders with consent from study participants.

ELIGIBILITY:
Inclusion Criteria:

* Aged 15 to 19 (Nigeria) and 15-24 (Ethiopia)
* Married
* Resident in a study geography
* For pregnant AGYW she should be at most 24 weeks gestation
* If not pregnant, AGYW should be at risk of pregnancy (not using a contraceptive method at the time of the survey with or without intend to conceive)

Exclusion Criteria:

* Married AGYW, aged 15-19 (Nigeria) or 15-24 (Ethiopia) who decline to give consent
* If pregnant, has an advanced pregnancy (≥ 25 weeks' gestation)
* If not pregnant, currently using a contraceptive method

Ages: 15 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2338 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Comprehensive knowledge of what is needed to pursue a healthy pregnancy | 3 months
  The proportion of AGYW who have 'comprehensive' knowledge of what is needed at conception to attain a healthy pregnancy. It is estimated as a composite measure derived from a combination of questions assessing AGYW's knowledge about pre-conceptual behaviors (proper nutrition, screening tests and treatment for HIV and sexually transmitted infections, use of prenatal vitamins, and avoidance of harmful substances).

SECONDARY OUTCOMES:
Pre-conceptual self-efficacy | 3 months
  The average item scores from a seven-item likert scale with five response options (strongly disagree=1 and strongly agree=5) administered to pregnant AGYW at recruitment and repeated after 3 months
Satisfaction of the support received from husband during pregnancy | 3 months
  The proportion of pregnant AGYW who are satisfied with the support they receive from husband during pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Population Services International, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: Yes
We are committed to ensuring that data from this study is available to other scientists for additional analysis. This in in line with the A360 donors' open access policy, encouraging scientists to deposit de-identified datasets on credible data repositories. We will therefore be availing de-identified datasets in recommended databases when the time comes.
Supporting Information: Study Protocol, ICF

DOCUMENTS (1):
  • Study Protocol (2024-08-22): https://cdn.clinicaltrials.gov/large-docs/65/NCT06680765/Prot_000.pdf